CLINICAL TRIAL: NCT04372940
Title: The Role of Tranexamic Acid in Aesthetic and Reconstructive Surgery
Brief Title: Tranexamic Acid in Gender Mastectomy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: due to COVID
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2019-0410-GM; A539730 (Other: UW Madison); SMPH/SURGERY/DENTL-PLASTC SRGY (Other: UW Madison)
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Surgery
Keywords: gender mastectomy; top surgery

STUDY DESIGN:
Intervention Model Description: TXA would be randomized to one side with the other acting as a control
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Side: TXA Irrigation (Experimental): 2.5% tranexamic acid will be applied directly to the wound via bulb irrigation and left in place for 5 minutes in the wound bed
  Interventions: Drug: Tranexamic Acid Irrigation
- Control Side: Saline Irrigation (Placebo Comparator): Contralateral side will serve as a control
  Interventions: Other: Saline Irrigation

INTERVENTIONS:
Drug: Tranexamic Acid Irrigation — Tranexamic acid (TXA) is a synthetic lysine analogue that inhibits the activation of plasminogen to plasmin, temporarily inhibiting the degradation of fibrin clots.
  Other Names: TXA
  Arms: Intervention Side: TXA Irrigation
Other: Saline Irrigation — Saline will serve as the control.
  Arms: Control Side: Saline Irrigation

SUMMARY:
The goal of this study is to examine the use of tranexamic acid (TXA) in gender mastectomy surgery, specifically looking at volume loss (blood and transudate) postoperatively.

DETAILED DESCRIPTION:
Anecdotal data from plastic surgeons around the country suggests that tranexamic acid has decreased patient's drain outputs, swelling, and bruising. Based on these anecdotal reports, many University of Wisconsin (UW) surgeons in Plastic and Reconstructive Surgery became interested in its use. It has a very safe profile and is inexpensive; therefore, many UW plastic surgeons have started using it topically prior to closure in many of procedures. Surgeons notice decreased drain output and bruising; and therefore decided to formally study the effects of tranexamic acid to determine whether there was a statistical difference in outcomes with the use of the drug.

For this sub-study, topical TXA will be applied to the surface of surgical sites and the primary outcome will be days to drain removal postoperatively. Secondary outcomes that would be assessed is total drain fluid output in milliliters, hematoma and seroma rates, and need for transfusion for hemoglobin < 7.0 postoperatively.

The hypothesis is that the use of TXA will result in earlier removal of drains by decreasing total drain fluid output and decreased need for transfusions, thus minimizing the associated complications/risks with drains and transfusions. The overall study is in two-parts, 1) a prospective study with retrospective controls via chart review and 2) a prospective controlled trial in bilateral procedures where participants serve as their own control with one side having tranexamic acid irrigation and the other side having saline irrigation.

This record documents a prospective controlled trial of the use of TXA in gender mastectomy, specifically.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing gender mastectomy
* English speaking

Exclusion Criteria:

* History of thrombotic event (ie deep vein thrombosis, pulmonary embolism, stroke, myocardial infarction)
* genetic disorder that increases risk of thrombosis
* use of estrogens at time of surgery
* pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — transgender males
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Days until drain removal | up to 30 days post-op

SECONDARY OUTCOMES:
Total drain output in mL for total time drain is in place | up to 30 days post-op
Drain fluid output in mL/day | up to 30 days post-op
Number of hematomas requiring aspiration or return to the operating room in the 30 days following surgery | up to 30 days post-op
Amount of fluid evacuated (mL) - hematomas | up to 30 days post-op
  Amount of fluid evacuated (mL) if hematomas require aspiration or return to the operating room in the 30 days following surgery
Number of seromas requiring aspiration or return to the operating room in the 30 days following surgery | up to 30 days post-op
Amount of fluid evacuated (mL) - seromas | up to 30 days post-op
  Amount of fluid evacuated (mL) if seromas require aspiration or return to the operating room in the 30 days following surgery
Number of Participants requiring transfusion for hemoglobin (Hgb) < 7.0 during postoperative admission | up to 30 days post-op
Number of units of blood transfused to maintain Hgb >7.0 in the postoperative admission | up to 30 days post-op

CONTACTS AND LOCATIONS:
Overall Officials: Katy Gast, MD, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No